CLINICAL TRIAL: NCT00182741
Title: Phase II Study of DN-101 (High Dose Pulse Calcitriol), Mitoxantrone, Prednisone in Androgen-Independent Prostate Cancer (AIPC)
Brief Title: Calcitriol, Mitoxantrone, and Prednisone in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Ryan, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441172; OHSU-8451; OHSU-VA-IRB-9451
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Mitoxantrone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: mitoxantrone hydrochloride
Drug: prednisone

SUMMARY:
RATIONALE: Calcitriol may cause prostate cancer cells to look more like normal cells, and to grow and spread more slowly. Drugs used in chemotherapy, such as mitoxantrone and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well giving calcitriol together with mitoxantrone and prednisone works in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the prostate-specific antigen (PSA) response rate, defined as the fraction of patients with 50% reduction in PSA level over 3 weeks' time, in patients with androgen-independent metastatic prostate cancer treated with high-dose pulse calcitriol, mitoxantrone, and prednisone.

Secondary

* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral high dose pulse calcitriol on day 1, mitoxantrone IV on day 2, and oral prednisone on days 1-21. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Androgen-independent disease, defined as disease progression while on standard hormonal management, including antiandrogen withdrawal

    * Patients must continue primary hormonal therapy during study treatment
  * Regional or distant metastases
* Prostate-specific antigen > 5 ng/mL
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 100

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Adequate hematologic function

Hepatic

* Adequate hepatic function

Renal

* Adequate renal function
* No calcium-salt kidney stones within the past 5 years
* No hypercalcemia

Cardiovascular

* Adequate cardiac function
* No significant cardiac disease
* No atrial fibrillation

Other

* Fertile patients must use effective barrier contraception during and for 2 months after completion of study treatment
* No other serious medical illness
* No other active malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* No prior strontium chloride Sr 89
* More than 28 days since prior radiotherapy
* More than 56 days since prior samarium Sm 153 lexidronam pentasodium

Surgery

* Prior prostatectomy and/or orchiectomy allowed

Other

* More than 28 days since prior investigational therapy

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Reduction in serum prostate-specific antigen (PSA) by 50% measured every 21 days

SECONDARY OUTCOMES:
Toxicity as measured by Common Toxicity Criteria v3.0
Frozen plasma and serum samples for correlative biomarker analysis collected every 21 days
Confirmed PSA reduction > 75% measured every 21 days
PSA normalization (< 4 ng/mL) measured every 21 days
Response to measurable disease as measured by RECIST criteria every 9 weeks
Analgesic response as measured by McGill-Melzack Pain Questionnaire every 21 days
Analgesic medication use decreased by ≥ 50% without an increase in pain for 2 consecutive evaluations at least 3 weeks apart
Palliative response as measured by McGill-Melzack Pain Questionnaire every 21 days
Quality of life as measured by EORTC core questionnaire Quality of Life-C30 every 21 days
Time to palliative-progression as measured by McGill-Melzack Pain Questionnaire every 21 days
Time to PSA progression measured every 21 days
Time to progression in measurable or evaluable disease as measured by whole body scan and/or CT or MRI scan every 9-12 weeks
Time to death assessed every 6 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. Ryan, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Chan JS, Beer TM, Quinn DI, Pinski JK, Garzotto M, Sokoloff M, Dehaze DR, Ryan CW. A phase II study of high-dose calcitriol combined with mitoxantrone and prednisone for androgen-independent prostate cancer. BJU Int. 2008 Dec;102(11):1601-6. doi: 10.1111/j.1464-410X.2008.08017.x. Epub 2008 Sep 8. PMID 18782306